CLINICAL TRIAL: NCT06865456
Title: Predictors of Survival of DKD Patients in Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hasnaa Osama Hassan Reiad, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: DKD predictors
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: diabetic nephropathy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: diapetic patient with diabetic nephropathy stage 4,5

SUMMARY:
In recent years, the global prevalence of diabetes has risen significantly. According to the 9th edition of the International Diabetes Federation Atlas, an estimated 463 million adults were living with diabetes in 2019, representing approximately 9.3% of the population, with an average annual increase of 51%.

Diabetes is associated with multiple complications that can significantly impact patient outcomes . In 2019 alone, around 4.2 million deaths were attributed to diabetes and its complications, accounting for approximately 11.3% of all global deaths .

In diabetic patients, several factors influence renal survival, including glycemic control, blood pressure management, lifestyle interventions, and pharmacological therapies such as renin-angiotensin-aldosterone system (RAAS) inhibitors, sodium-glucose co-transporter-2 (SGLT2) inhibitors, and glucagon-like peptide-1 (GLP-1) receptor agonists(9). Early detection of kidney dysfunction through biomarkers like estimated glomerular filtration rate (eGFR) and urinary albumin-to-creatinine ratio (UACR) plays a pivotal role in improving renal outcomes.

This study aims to evaluate the factors affecting Patients survival in diabetic patients, identify early predictors of renal function decline, and assess the effectiveness of current therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* ● Patients age > 18 years old

  * Both sex
  * diabetic patients with HbA1c level >6.5( Type 1 and 2)
  * Diabetic patients with CKD 4, 5 )
  * HD Pt

Exclusion Criteria:

* ● Chronic kidney diseases stage 1,2, and 3.

  * Acute kidney injury.
  * Patients with any other causes of CKD autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diabetic patients with chronic kideny disease stage 4,5
Sampling Method: Probability Sample
Enrollment: 129 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
incidence of CKD in diabetic patients | baseline
  pergentage of diabetic patients with stage 4,5 chronic kidney disease